CLINICAL TRIAL: NCT04747392
Title: A Randomized, Open, Self-crossover, Single-dose Clinical Study to Compare Pharmacokinetic of Teriparatide Injection (SAL001) and the Original Drug FORSTEO in Healthy Chinese Adult Volunteers
Brief Title: Bioequivalence Study of SAL001 and FORSTEO in Healthy Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAL001A101
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Teriparatide; Bioequivalence
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Other): The test drug (SAL001) is administrated once by subcutaneous injection in the first period, and the reference drug (FORSTEO) is administrated once by subcutaneous injection in the second period.
  Interventions: Biological: SAL001; Biological: FORSTEO
- Sequence B (Other): The reference drug (FORSTEO) is administrated once by subcutaneous injection in the first period, and the test drug (SAL001) is administrated once by subcutaneous injection in the second period.
  Interventions: Biological: SAL001; Biological: FORSTEO

INTERVENTIONS:
Biological: SAL001 — administrated once by subcutaneous injection
Biological: FORSTEO — administrated once by subcutaneous injection

SUMMARY:
This is a single-center, randomized, open label, single-dose, the original drug controlled, crossover design, two sequence, two periods, Phase Ⅰclinical study.

64 qualified subjects will be randomly assigned to two administration sequences (sequence A and sequence B) at the ratio of 1∶1, with 32 subjects in each sequence. Each period will be given subcutaneous injection once, and the washout period will be 72 hours, and each subject will be given subcutaneous injection twice. Sequence A: the test drug (SAL001) is injected in the first period, and the reference drug (FORSTEO) is injected in the second period. Sequence B: the reference drug (FORSTEO) is injected in the first period, and the test drug (SAL001) is injected in the second period.

If the geometric mean ratio (GMR) 90% confidence interval of the major pharmacokinetic indexes (AUC0-t, Cmax) for SAL001 and FORSTEO is between 80.00% and 125.00%, the two drugs are considered to be bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

1. Those who volunteer to participate in the trial and sign the informed consent form.
2. Healthy Chinese male or female adults, the number of single sex volunteers is no less than 1/3, aged 20 to 50 years old (including the boundary value).
3. Males weighted ≥50kg, females weighted ≥45kg, body mass index (BMI) between 19-25 kg/m^2 (including boundary value), BMI= weight (kg)/height^2 (m^2).

Exclusion Criteria:

1. The existence of clinically significant diseases of heart, liver, lung, kidney, digestive tract, endocrine, metabolic and hematological systems.
2. history of parathyroid disease, or abnormal PTH with clinically significance judged by investigators.
3. Physical examination, laboratory examination, electrocardiogram (ECG), chest radiograph, abdominal ultrasound san(digestive system, urinary system), vital signs, etc., indicate that the subject has clinically significant abnormalities judged by the investigator.
4. Serum total calcium > upper limit of normal according to the normal range of the center, or previous hypercalcemia.
5. Hyperuricemia, or a previous history of gout, or abnormal blood uric acid with clinically significance judged by investigators at the time of screening.
6. Those with active urolithiasis.
7. Those who had received anti-osteoporosis agents (such as bisphosphonates, calcitonin, estrogen, selective estrogen receptor modulator, parathyroid hormone and its analogues, strontium salts, active vitamin D and its analogues, vitamin K2, etc.) within 6 months before the first administration of the trial.
8. Those who had received oral or intravenous administration of glucocorticoids 3 months before the first administration of the trial.
9. Those who had taken any drug within 14 days before the first administration of the trial.
10. Allergies, such as allergic to two or more kinds of drugs or food; or known allergic to this drug components.
11. Alcoholism within 1 year before screening (drinking more than 3 times a day or more than 7 times a week, drinking 1 time =150mL red wine, or 360mL beer, or 50mL white wine), or a positive alcohol breath test.
12. A history of drug abuse within 1 year before screening, or a positive urine test for drugs at screening.
13. Those who were smoking more than 5 cigarettes a day within 3 months before screening.
14. Those who had participated in any other clinical trial within 3 months before the first administration of the trial.
15. Those who had blood donation or blood loss ≥400mL within 3 months before the first administration of the trial.
16. Those who do not agree to avoid the use of tobacco, alcohol or caffeinated beverages within 24 hours before the administration and during the trial, or do not agree to avoid strenuous exercise, or do not agree to avoid other factors affecting the absorption, distribution, metabolism and excretion of the drug.
17. Women who are pregnant or lactating, or who are positive for serum HCG, or who cannot/do not follow the instructions of investigators to take contraceptive measures approved by investigators during the study period.
18. Those who intend to give birth within 1 year.
19. Those with positive results of HBV surface antigen, or hepatitis C virus antibody positive, or Treponema pallidum antibody positive, or human immunodeficiency virus antibody positive.
20. Those with positive results of novel coronavirus nucleic acid test.
21. Those who are considered to be unsuitable for participation in this clinical study by investigators.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
PK parameters: area under the plasma concentration time curve from-time zero to time t (AUC0-t) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: peak plasma concentration (Cmax) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.

SECONDARY OUTCOMES:
PK parameters: area under the plasma concentration time curve from time zero to time infinity (AUC0-∞) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: time to reach peak drug concentration (Tmax) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: half-life (t1/2) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: AUC extrapolated from Tmax to infinity in percentage of the total AUC (AUC%extrap) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: time to last measurable concentration (Tlast) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: terminal elimination rate constant (λz) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: apparent total clearance (CL/F) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: apparent distribution volume (Vz/F) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: mean residence time from time zero to t (MRT0-t) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PK parameters: mean residence time from time zero to infinity (MRT0-∞) | Within 60 minutes before administration, and 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 210, 240, and 300 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the plasma concentration of drugs.
PD parameters: area under the serum concentration time curve from-time zero to time t (AUC0-t) | Within 60 minutes before administration, and 120, 180, 240, 360, 480, 720 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the serum total calcium concentration. Serum-corrected calcium concentration will be use to calculate above PD parameters.
PD parameters: area under the serum concentration time curve from time zero to time infinity (AUC0-∞) | Within 60 minutes before administration, and 120, 180, 240, 360, 480, 720 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the serum total calcium concentration. Serum-corrected calcium concentration will be use to calculate above PD parameters.
PD parameters: peak serum concentration (Cmax) | Within 60 minutes before administration, and 120, 180, 240, 360, 480, 720 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the serum total calcium concentration. Serum-corrected calcium concentration will be use to calculate above PD parameters.
PD parameters: time to reach peak serum concentration (Tmax) | Within 60 minutes before administration, and 120, 180, 240, 360, 480, 720 minutes after administration of Day 1 and Day 4
  Central lab will be used to detect the serum total calcium concentration. Serum-corrected calcium concentration will be use to calculate above PD parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No